CLINICAL TRIAL: NCT06572605
Title: A Phase 1b/2 Study of Talquetamab Plus Concomitant Priming Radiotherapy in Multiple Myeloma With Extramedullary Disease
Brief Title: External Beam Radiation Therapy in Combination With Talquetamab for the Treatment of Multiple Myeloma Patients With Extramedullary Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23931; NCI-2024-06707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23931 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Extramedullary Disease in Multiple Myeloma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; Congresses as Topic; Radiation; Image-Guided Biopsy; X-Rays; Magnetic Resonance Spectroscopy; talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (EDM-EBRT, talquetamab) (Experimental): STEP-UP PERIOD: Patients undergo EMD-EBRT QD for 5 treatment fractions on weekdays (Monday to Friday), and receive talquetamab SC starting after the first fraction of EMD-EBRT and continuing every 2-4 days for up to 3 step-up doses in the absence of unacceptable toxicity.
  SUBSEQUENT TREATMENT: Starting 2-7 days after step-up dose 3, patients receive talquetamab SC on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to a maximum of 13 total cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT and/or PET/CT and collection of blood samples throughout the trial and undergo image-guided EMD biopsy at screening and on study. Patients undergo bone marrow biopsy/aspiration at screening and optionally at end of treatment.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Electronic Health Record Review; Radiation: External Beam Radiation Therapy; Procedure: Image Guided Biopsy; Procedure: Positron Emission Tomography; Biological: Talquetamab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Radiation: External Beam Radiation Therapy — Undergo EMD-EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: Image Guided Biopsy — Undergo image-guided EMD biopsy
  Other Names: Image-Guided Biopsy; Imaging for Biopsy; Imaging Guided Biopsy
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Talquetamab — Given SC
  Other Names: Anti-CD3/Anti-GPRC5D Bispecific Monoclonal Antibody JNJ-64407564; GPRC5D x CD3 Bispecific Antibody JNJ-64407564; GPRC5D x CD3 DuoBody Antibody JNJ-64407564; GPRC5D/CD3 DuoBody Antibody JNJ-64407564; Humanized GPRC5D x CD3 DuoBody Antibody JNJ-64407564; JNJ 64407564; JNJ-64407564; JNJ64407564; Talquetamab-tgvs

SUMMARY:
This phase I/II trial tests the safety and effectiveness of extramedullary disease (EMD)-directed external beam radiation therapy (EBRT) in combination with talquetamab for the treatment of multiple myeloma patients with extramedullary disease. Extramedullary disease in multiple myeloma involves the infiltration of organs and soft tissues by malignant plasma cells and has proven difficult to treat. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink cancers. EBRT is a type of radiation therapy that delivers high-energy beams to the cancer from outside of the body. In this trial, the EBRT will be directed to a site of extramedullary disease. Talquetamab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Combining EMD-directed EBRT with talquetamab may be safe, tolerable, and/or effective in treating multiple myeloma patients with extramedullary disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of single-field, palliative, extramedullary disease (EMD)-directed external beam radiotherapy (EMD-EBRT) in combination with talquetamab as assessed by incidence of adverse events (AEs) throughout the trial and unexpected toxicities (UTs) during step-up and cycle 1. (Phase 1b) II. To evaluate the systemic anti-tumor activity/preliminary efficacy of EMD-EBRT in combination with talquetamab as assessed by EMD-modified overall response rate (ORR). (Phase 2)

SECONDARY OBJECTIVE:

I. To additionally evaluate efficacy through International Myeloma Working Group (IMWG) overall response rate (ORR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To assess the impact of EMD-EBRT combined with talquetamab on peripheral blood immune cell populations.

II. To assess the spatial transcriptomic changes in the medullary and extramedullary tumor microenvironment in response to EMD-EBRT combined with talquetamab.

OUTLINE:

STEP-UP PERIOD: Patients undergo EMD-EBRT once daily (QD) for 5 treatment fractions on weekdays (Monday to Friday), and receive talquetamab subcutaneously (SC) starting after the first fraction of EMD-EBRT and continuing every 2-4 days for up to 3 step-up doses in the absence of unacceptable toxicity.

SUBSEQUENT TREATMENT: Starting 2-7 days after step-up dose 3, patients receive talquetamab SC on days 1 and 15 of each cycle. Cycles repeat every 28 days for up to a maximum of 13 total cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo computed tomography (CT) and/or positron emission tomography (PET)/CT and collection of blood samples throughout the trial and undergo image-guided EMD biopsy at screening and on study. Patients undergo bone marrow biopsy/aspiration at screening and optionally at end of treatment.

After completion of study treatment, patients are followed up every 28 days for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Karnofsky performance status (KPS) ≥ 60%
* Diagnosis of multiple myeloma with extramedullary disease (EMD). EMD is defined as soft-tissue plasmacytomas NOT arising from skeletal lesions (i.e., the EMD is not contiguous with any bone/bony lesion)
* Measurable systemic disease defined as serum M-spike ≥ 0.5 g/dl, 24-hour urine M-spike ≥ 200 mg/24 hours (hr), involved serum free light chain (FLC) ≥ 10 mg/dl with abnormal FLC ratio, and/or a non-target plasmacytoma ≥ 2 cm in a single diameter (NOTE: Non-target plasmacytoma must not be included in the EMD-EBRT field)
* At least one site of EMD must have an indication for palliative radiation per the treating clinicians (e.g., including but not limited to pain, asymmetry, discomfort, threatening to vital structure, etc.)
* Target EMD site must be encompassed by one radiation field per treating radiation oncologist
* Subject must have received an immunomodulatory agent, a proteasome inhibitor, and an anti-CD38 antibody
* Fully recovered from the acute non-hematologic toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Prior antitumor therapy must have been completed prior to enrollment as follows:

  * ≥ 2 weeks for prior external beam radiotherapy (XRT) to non-target site
  * ≥ 21 days for cytotoxic chemotherapy (systemic or intrathecal)
  * ≥ 28 days for prior adoptive cell therapy or T-cell redirecting therapies
  * ≥ 4 weeks or 5 half-lives (whichever is shorter) for other myeloma therapies
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (prior growth factor support is permitted but must be without support for 7 days for granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM-CSF] and for 14 days for pegylated GCSF before the laboratory test)

  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Platelets ≥ 50,000/mm^3

  * NOTE: No transfusion support or thrombopoietin receptor agonist within 7 days before laboratory test
  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Hemoglobin ≥ 8g/dL

  * NOTE: No transfusion support or erythropoietin use within 7 days before the laboratory test
  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Total bilirubin ≤ 2.0 X upper limit of normal (ULN) (unless has congenital bilirubinemia such as Gilbert's disease, in which case ≤ 1.5 × ULN is required)

  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN

  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN

  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Creatinine clearance of ≥ 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula

  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Two repeat tests are allowed. If the repeat test satisfies criteria, the participant may enroll provided all other criteria are met
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of talquetamab

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior irradiation to target EMD site or field
* Prior GPRC5D therapy
* Prior radiopharmaceutical therapy
* Patients who have received previous radiation to > 25% of their bone marrow
* Prior allogeneic hematopoietic cell transplantation within the past 6 months or prior autologous hematopoietic cell transplantation within the past 12 weeks
* A maximum cumulative dose of corticosteroids of ≥ 140 mg of prednisone or equivalent within 14-day period before the first dose of study drug (does not include pre-treatment medications)
* Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study, or within 2 weeks after administration of the last dose of study treatment

  * Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the investigator must consult with the appropriate representative at Janssen and resolve any issues before enrolling a participant in the study
* Ongoing or active infection
* Severe persistent asthma or severe chronic obstructive pulmonary disease (COPD)
* Presence of the following cardiac conditions:

  * New York Heart Association stage III or IV congestive heart failure
  * Myocardial infarction or coronary artery bypass graft ≤ 6 months prior to randomization
  * Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  * History of severe non-ischemic cardiomyopathy
* Any of the following:

  * Hepatitis B infection (i.e., hepatitis B virus surface antigen [HBsAg] or hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status
  * Active hepatitis C infection as measured by positive hepatitis C virus [HCV]-ribonucleic acid [RNA] testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA for at least 12 weeks following the completion of therapy, the participant is eligible for the study
* Plasma cell leukemia (> 20% circulating plasma cells and/or > 2.0 x 10^9/L plasma cells) at the time of screening, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary amyloid light chain amyloidosis
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Stroke or seizure within 6 months prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* If HIV positive, any of the following:

  * Detectable viral load at screening
  * CD4+ T cell count ≤ 300
  * AIDS-defining opportunistic infection within 6 months of screening
  * Changes in highly active antiretroviral therapy (HAART) due to resistance/progression that occurred within 3 months prior to screening
  * Changes in HAART due to toxicity within 4 weeks prior to screening
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2030-01-18 (Estimated); Study Completion 2030-01-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (phase 1b) | From start of protocol therapy until cycle 1 day 28
  Toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome. Toxicity information recorded in each patient will include the type, severity, and the probable association with the study regimen. Tabular and graphical summaries will be used to represent the observed incidence by severity and type of toxicity.
Extramedullary disease (EMD)-modified overall response rate (ORR) (phase 2) | Up to 12 months
  EMD-modified ORR will be defined as the proportion of patients meeting the criteria for partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR). Disease response will be evaluated per International Myeloma Working Group (IMWG) response criteria and Response Criteria for EMD. Clopper-Pearson 95% confidence intervals will be calculated for these estimates.

SECONDARY OUTCOMES:
Progression-free survival | From first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 12 months
  Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival | From first day of treatment to time of death due to any cause, assessed up to 12 months
  Will be estimated using the product-limit method of Kaplan and Meier.
Duration of response | From first response documented until disease progression, assessed up to 12 months
  Will be evaluated in patients with PR or better. Will be estimated using the product-limit method of Kaplan and Meier.
Clinical benefit rate | Up to 12 months
  Clinical benefit rate will be defined as the proportion of patients meeting the criteria for stable disease, PR, VGPR, CR, or sCR. Disease response will be evaluated per IMWG response criteria. Clopper-Pearson 95% confidence intervals will be calculated for these estimates.
Incidence of adverse events | Up to 12 months
  Will evaluate the frequency and severity of adverse events, severe adverse events, laboratory abnormalities. Toxicity information recorded in each patient will include the type, severity, and the probable association with the study regimen. Tabular and graphical summaries will be used to represent the observed incidence by severity and type of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Goldsmith, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States